CLINICAL TRIAL: NCT01615991
Title: Multicentre Canadian Study to Measure the Safety and Efficacy of Synoviorthesis Performed With Yttrium-90 or Rhenium-186 Sulfide
Brief Title: Multicentre Canadian Study to Measure the Safety and Efficacy of Radiosynoviorthesis
Acronym: RSO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Principal Investigator, Dr Éric E Turcotte, MD, Head, Clinical research, Centre d'imagerie moléculaire de Sherbrooke; Associate Professor, Université de Sherbrooke;Nuclear Medecine Specialist, Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIMS-2012-01
Record Dates: First submitted 2012-05-14; First posted 2012-06-11 (Estimated); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- radiosynoviorthesis with yttrium-90 or rhenium -186 (Other): Patients suffering from arthritis or chronic inflammatory joint disease.
  Interventions: Drug: Radiosynoviorthesis

INTERVENTIONS:
Drug: Radiosynoviorthesis — Intraarticular administration from 111 to 222 Mbq yttrium-90 per joint
  Other Names: Yttrium-90 colloid suspension for local injection

SUMMARY:
Radiation synovectomy by intra-articular injection of beta-emitting radionuclides is considered a reliable and easy-to-perform therapy without harmful side-effects for the treatment of inflammatory joint disease in many countries.

The goal of this study is to demonstrate Yttrium-90 citrate colloid or Rhenium-186 sulfide synovectomy are appropriate therapeutic interventions in patients with persistent active synovitis of a joint (characterized by pain, tenderness, and effusion) which is resistant to systemic therapy and intra-articular corticosteroid injections.

The primary objective will be to assess the safety of an intra-articular administration of Yttrium-90 citrate colloid or Rhenium-186 sulfide.

The secondary objective will be to assess the efficacy on synovitis.

ELIGIBILITY:
Inclusion Criteria:

* There is no age limit for RSO
* Patient referred by a medical joint specialist (orthopedist, rheumatologist or internal medicine in the absence of local joint specialist)
* Patient having a refractory inflammatory articular disease:
* Failure of medical therapy after 6 months
* Clinical signs of an active mono or oligo synovitis
* Joint X-ray, echo or MR showing minimal cartilage or bone destruction
* Pain limits normal activities or requires significant analgesic medication

Exclusion Criteria:

* Prior RSO within last 3 months in that joint
* Collapse of the articular plateau or intra-articular fracture
* Surgery or arthroscopy within last 6 weeks
* Painful prosthesis
* Joint infection, local skin infection, bacteremia
* Joint puncture within last 2 weeks (increased risk of soft tissue necrosis along the needle track)
* Pregnancy or breast feeding
* Synovial cyst rupture
* Massive hemarthrosis
* Generalized synovitis defined as more than 5 uncontrolled joints by clinical examination or 3 phases bone scan
* Surgical synovectomy within 6months
* Cancer with bone metastases
* Hypersensitivity, allergies or contraindication to the used radiopharmaceutical agent
* Participation in any other ongoing clinical trial for the underlying inflammatory condition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-05-31; Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
safety | 3-4 days post -treatment
  The safety profile will be assessed by the incidence of AEs. All the AEs will be described by system/organ class and preferred terms and overall sorted by frequency.

SECONDARY OUTCOMES:
Efficacy | Clinical response post treatment
  Efficacy outcomes will be the clinical response over 1 year post treatment ( at 3, 6 and 12 months):The comparison will be done with a confidence interval approach based on a Chi²-test for each of the above secondary criterion assessed at different times during the follow-up compared to the same criterion assessed at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Turcotte, MD, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (9):
- Canada (9):
  - Alberta Children's Hospital, Calgary, Alberta
  - Lion's Gate Hospital, Vancouver, British Columbia
  - Health Science Centre, Winnipeg, Manitoba
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Centre de santé et services sociaux Pierre-Boucher, Hôpital Pierre-Boucher, Longueuil, Quebec
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - CHR Trois-Rivières, Trois-Rivières, Quebec
  - Centre Hospitalier Universitaire de Québec, Québec